CLINICAL TRIAL: NCT06705972
Title: Comparing the Accuracy of Different Ultrasound -based Scores to Assess Disease Severity in Patients with Inflammatory Bowel Disease
Brief Title: Comparing the Accuracy of Different Ultrasound-based Scores to Assess Disease Severity in Patients with Inflammatory Bowel Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martina Mamdouh Zekry Ayoub, Resident, Assiut University
Other Study IDs: Role of ultrasound in IBD
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: inflammatory bowel disease,ultrasound,scoring
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Infammatory Bowel Disease (IBD) is a lifelong chronic disease comprised of two main entities: Crohn's disease and Ulcerative Colitis. The former can involve any part of the gastrointestinal tract with marked mural infammatory change and frequent complications related to either a penetrating or fbrostenotic phenotype, while the latter is a superfcial inflammatory process involving only the colon. IBD can undergo spontaneous periods of remission and activity and has a full spectrum from mild inconsequential disease to incapacitating complications, which may alter both lifestyle and longevity The aim of research is to compare between different ultrasound based scores used to assess disease severity in patients with inflammatory bowel disease to determine the most accurate score to be validated to use in clinical practice

DETAILED DESCRIPTION:
* Infammatory Bowel Disease (IBD) is a lifelong chronic disease comprised of two main entities: Crohn's disease and Ulcerative Colitis. The former can involve any part of the gastrointestinal tract with marked mural infammatory change and frequent complications related to either a penetrating or fbrostenotic phenotype, while the latter is a superfcial inflammatory process involving only the colon. IBD can undergo spontaneous periods of remission and activity and has a full spectrum from mild inconsequential disease to incapacitating complications, which may alter both lifestyle and longevity
* IBD patients require repeat imaging throughout the course of their disease, necessitating a safe, noninvasive, available, and repeatable method. Imaging is required at diagnosis, routine surveillance, and acute flare of disease. Ultrasound imaging meets these demands with a high degree of accuracy and wide patient acceptance. Ultrasound provides high-resolution imaging and is excellent for detailed evaluation of the bowel wall and surrounding soft tissues performed without ionizing radiation with an extremely low risk of adverse contrast events compared to CT and MR Enterography which use ahigh dose of ionizing radiation, making it the frst choice of many Gastroenterologists and overwhelmingly preferred by patients

Several established IUS parameters are assessed during an IUS examination. These include bowel wall thickness (BWT); the stratification of the bowel wall layers, blood flow, luminal diameters, and motility, Additional extraintestinal surrogates to bowel inflammation to assess for include mesenteric fat proliferation and lymphadenopathy ,with proposal of different sonographic scoring systems in this domain to predict disease severity

ELIGIBILITY:
Inclusion Criteria:

- Adult patients aged 18-70 Confirmed diagnosis of Crohn's Disease or Ulcerative Colitis based on clinical, endoscopic, and histologic criteria

Exclusion Criteria:

* Patients with other gastrointestinal diseases History of colectomy or proctocolectomy: Patients without a colon or rectum, which would limit the ability to assess IBD in those regions using ultrasound

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample size was calculated using the sample size calculator for sensitivity and specificity studies described by Dr Lin Naing @ Mohd. Ayub Sadiq (School of Dental Sciences, Universiti Sains Malaysia, Penang, Malaysia). Based on determining the main outcome variabble which is To compare the efficacy of different ultrasound scoring systems in assessing disease severity in IBD patients and To determine the correlation between ultrasound scores and clinical, endoscopic, and histological findings According to the following inputs: expected sensitivity of the ultrasound in detecting IBD patients = 92%, expected Specificity =75%,*(9)* , desired precision = 6%, Confidence level = 80%. Sample size was 60 cases.Sample size was calculated using the sample size calculator for sensitivity and specificity studies described
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To compare efficacy of different ultrasound scores to assess disease severity in IBD patients | Baseline
  To compare the efficacy of different ultrasound scoring systems in assessing disease severity in IBD patients.
  To determine the correlation between ultrasound scores and clinical, endoscopic, and histological findings
  .To identify the most reliable and practical ultrasound scoring system for routine clinical use

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rimola J, Torres J, Kumar S, Taylor SA, Kucharzik T. Recent advances in clinical practice: advances in cross-sectional imaging in inflammatory bowel disease. Gut. 2022 Dec;71(12):2587-2597. doi: 10.1136/gutjnl-2021-326562. Epub 2022 Aug 4. PMID 35927032
- [Background] Valette PJ, Rioux M, Pilleul F, Saurin JC, Fouque P, Henry L. Ultrasonography of chronic inflammatory bowel diseases. Eur Radiol. 2001;11(10):1859-66. doi: 10.1007/s003300101065. PMID 11702118
- [Background] Allocca M, Dell'Avalle C, Craviotto V, Furfaro F, Zilli A, D'Amico F, Bonovas S, Peyrin-Biroulet L, Fiorino G, Danese S. Predictive value of Milan ultrasound criteria in ulcerative colitis: A prospective observational cohort study. United European Gastroenterol J. 2022 Mar;10(2):190-197. doi: 10.1002/ueg2.12206. Epub 2022 Mar 1. PMID 35233934
- [Background] Dragoni G, Gottin M, Innocenti T, Lynch EN, Bagnoli S, Macri G, Bonanomi AG, Orlandini B, Rogai F, Milani S, Galli A, Milla M, Biagini MR. Correlation of Ultrasound Scores with Endoscopic Activity in Crohn's Disease: A Prospective Exploratory Study. J Crohns Colitis. 2023 Oct 20;17(9):1387-1394. doi: 10.1093/ecco-jcc/jjad068. PMID 37023010
- [Background] Goodsall TM, Nguyen TM, Parker CE, Ma C, Andrews JM, Jairath V, Bryant RV. Systematic Review: Gastrointestinal Ultrasound Scoring Indices for Inflammatory Bowel Disease. J Crohns Colitis. 2021 Jan 13;15(1):125-142. doi: 10.1093/ecco-jcc/jjaa129. PMID 32614386